CLINICAL TRIAL: NCT02893826
Title: Multicenter, Controlled, Randomized, Safety and Pharmacokinetic Study Comparing Intracisternal EG-1962 to Standard of Care Enteral Nimodipine in Adults With Aneurysmal Subarachnoid Hemorrhage
Brief Title: Safety/Pharmacokinetic Study Comparing Intracisternal EG-1962 to Standard of Care Enteral Nimodipine in Adults With aSAH
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on DMC recommendation to discontinue EG-01-1962-03
Sponsor: Edge Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EG-01-1962-04
Record Dates: First submitted 2016-08-25; First posted 2016-09-09 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: Aneurysm; Ruptured; nimodipine; subarachnoid hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage; Aneurysm; Rupture | interventions — EG-1962

ARMS (2):
- EG-1962 Group (Experimental): 1 dose of intracisternal EG-1962 (nimodipine microparticles) 600 mg
  Interventions: Drug: EG-1962 (nimodipine microparticles)
- Enteral Nimodipine Group (Active Comparator): Up to a total of 21 days of enteral nimodipine (including nimodipine received prior to randomization)
  Interventions: Drug: Enteral Nimodipine

INTERVENTIONS:
Drug: EG-1962 (nimodipine microparticles)
  Other Names: Single intracisternal adminstration
  Arms: EG-1962 Group
Drug: Enteral Nimodipine
  Other Names: Administered for up to 21 days
  Arms: Enteral Nimodipine Group

SUMMARY:
Safety and Pharmacokinetic study comparing intracisternal EG-1962 to enternal nimopidine in the treatment of aneurysmal subarachnoid hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

1. Ruptured saccular aneurysm repaired by neurosurgical clipping
2. Subarachnoid hemorrhage on computed tomography (CT) scan of grade 2-4 on the modified Fischer scale
3. WFNS grade 1 or 2 assessed during the Pre-randomization Phase. If WFNS grade 2, must not require an EVD prior to aneurysm repair

Exclusion Criteria:

1. Major complication during aneurysm repair such as, but not limited to, massive intraoperative hemorrhage, brain swelling, arterial occlusion or inability to secure the ruptured aneurysm
2. Angiographic vasospasm prior to randomization
3. Evidence of cerebral infarction with neurological deficit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-09; Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 90 Days
Proportion of subjects with delayed cerebral infarctions present on CT at Day 30 | 30 Days

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of EG-1962 as measured by maximum drug concentration in plasma (Cmax) | At the time of the first post-operation blood draw and every 6 hours (± 30 minutes) for the first 24 hours and daily thereafter until hospital discharge or Day 21, whichever occurs first and Day 30
Pharmacokinetic (PK) profile of EG-1962 as measured by time to reach maximum drug concentration in plasma (Tmax) | At the time of the first post-operation blood draw and every 6 hours (± 30 minutes) for the first 24 hours and daily thereafter until hospital discharge or Day 21, whichever occurs first and Day 30
Pharmacokinetic (PK) profile of EG-1962 as measured by steady state concentration (Css) | At the time of the first post-operation blood draw and every 6 hours (± 30 minutes) for the first 24 hours and daily thereafter until hospital discharge or Day 21, whichever occurs first and Day 30
Pharmacokinetic (PK) profile of EG-1962 as measured by AUC area under the plasma concentration-time curve (AUC) from 0 to 24 hours (AUC024h) | At the time of the first post-operation blood draw and every 6 hours (± 30 minutes) for the first 24 hours
Pharmacokinetic (PK) profile of EG-1962 as measured by AUC from 0 to Day 10 (AUC0-10) | At the time of the first post-operation blood draw and every 6 hours (± 30 minutes) for the first 24 hours and up to Day 10
Pharmacokinetic (PK) profile of EG-1962 as measured by AUC from 0 to Day 14 (AUC0-14) | At the time of the first post-operation blood draw and every 6 hours (± 30 minutes) for the first 24 hours and up to Day 14
Pharmacokinetic (PK) profile of EG-1962 as measured by AUC from 0 to last plasma concentration (AUC0-last) | At the time of the first post-operation blood draw and every 6 hours (± 30 minutes) for the first 24 hours and up to last plasma concentration

OTHER OUTCOMES:
Extended Glasgow Outcome Scale (GOSE) | Day 90
  Proportion of subjects with a favorable outcome measured on the Extended Glasgow Outcome Scale (GOSE) at Day 90
Montreal Cognitive Assessment (MoCA) | Day 90
  Proportion of subjects with a favorable outcome measured on the Montreal Cognitive Assessment (MoCA) at Day 90

CONTACTS AND LOCATIONS:
Overall Officials: R. Loch Macdonald, MD, PhD, Study Chair — Edge Therapeutics Inc
Locations (4):
- United States (3):
  - Dignity Health; St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of California San Francisco, San Francisco, California
  - University of Maryland Medical Systems, Baltimore, Maryland
- University of Alberta Hospital/Mackenzie Health Sciences Centre, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De BP, Rosenberg JB, Selvan N, Wilson I, Yusufzai N, Greco A, Kaminsky SM, Heier LA, Ricart Arbona RJ, Miranda IC, Monette S, Nair A, Khanna R, Crystal RG, Sondhi D. Assessment of Safety and Biodistribution of AAVrh.10hCLN2 Following Intracisternal Administration in Nonhuman Primates for the Treatment of CLN2 Batten Disease. Hum Gene Ther. 2023 Sep;34(17-18):905-916. doi: 10.1089/hum.2023.067. PMID 37624739
- [Derived] Macdonald RL, Hanggi D, Ko NU, Darsaut TE, Carlson AP, Wong GK, Etminan N, Mayer SA, Aldrich EF, Diringer MN, Ng D, Strange P, Bleck T, Grubb R, Suarez JI. NEWTON-2 Cisternal (Nimodipine Microparticles to Enhance Recovery While Reducing Toxicity After Subarachnoid Hemorrhage): A Phase 2, Multicenter, Randomized, Open-Label Safety Study of Intracisternal EG-1962 in Aneurysmal Subarachnoid Hemorrhage. Neurosurgery. 2020 Dec 15;88(1):E13-E26. doi: 10.1093/neuros/nyaa430. PMID 32985652